CLINICAL TRIAL: NCT07337629
Title: Comparison of the Effects of Single Dose Preemptive Paracetamol or Ibuprofen Administration Before Septrorhinoplasty on Intra- and Postoperative Opioid Consumption.
Brief Title: Single Dose Preemptive Paracetamol or Ibuprofen Before Septrorhinoplasty on Intra- and Postoperative Opioid Consumption.
Status: Recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK 2025/22/11
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Analgesia
Keywords: SEPTORHİNOPLASTY; PREEMPTİVE; PARACETEMOL; IBUPROFEN
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- GROUP P: PARACETEMOL
- GROUP I: IBUPROFEN
- GROUP K: CONTROL

SUMMARY:
Reducing intra- and postoperative pain or using less opioids is an essential strategy in today's operations. One emerging and widely used method in this context is the use of preemptive analgesic medication. Paracetamol and ibuprofen used preemptively have been shown to reduce postoperative opioid use and pain scores. There are also studies showing that preemptive analgesia with different analgesic medications reduces opioid consumption and postoperative pain. Our study will evaluate both the intraoperative and postoperative effectiveness of paracetamol and ibupurofen with preemptive analgesia, considering total opioid use. It will also investigate drug side effects and their advantages using a 15-question compilation quality scale, validated in Turkish.

DETAILED DESCRIPTION:
Our study will be prospective, observational, and conducted through face-to-face interviews with patients at the Ear, Nose, and Throat Operating Room, Anesthesiology and Reanimation Clinic of Samsun University, Samsun Training and Research Hospital. The study is planned to begin on November 1, 2025, and be completed by August 31, 2026. The study will be conducted by Dr. Hasan CETINKAYA and Dr. Hatice SELCUK KUSDERCI.

Sample size calculation for data analysis was based on data from a reference study (Alshehri AA, Int Arch Otorhinolaryngol. 2023;27(3):e471-e477) evaluating the effect of preemptive analgesic agents on opioid consumption after septorhinoplasty surgery. In the reference study, total opioid consumption (mg) was reported as mean ± standard deviation as 486.4 ± 40.84 mg in Group A, 410.2 ± 88.41 mg in Group B, and 372.8 ± 90.45 mg in Group C. The pooled standard deviation calculated from these values was 76.8 mg, and the Cohen's f effect size was obtained as 0.615 based on the differences between the group means. Using G*Power 3.1 software, a priori power analysis was performed for one-way ANOVA (one-way fixed effects omnibus) with parameters α = 0.05, power (1-β) = 0.95, and number of groups = 3. The minimum total sample size was calculated as 45 (15 participants per group). In our study, the planned sample size was increased to compensate for potential losses and omissions. This aimed to achieve the expected effect size (f = 0.615) and 95% statistical power at the determined significance level.

Statistical analysis: The data obtained in the research will be analyzed using IBM SPSS Statistics (version 25.0 or higher) software. All data will first be summarized with descriptive statistics, expressing mean ± standard deviation or median (min-max) values for continuous variables, and number and percentage (%) for categorical variables. The distribution characteristics of the data will be evaluated using the Shapiro-Wilk test for intergroup comparisons. One-way analysis of variance (ANOVA) will be used for continuous variables showing a normal distribution; when a significant difference is found, the Tukey HSD post-hoc test will be applied for intragroup pairwise comparisons. For variables not showing a normal distribution, the Kruskal-Wallis test will be preferred; when a difference is found, pairwise comparisons will be made using the Mann-Whitney U test with Dunn-Bonferroni correction. Differences between categorical variables will be evaluated using the Chi-square test (χ²) or, if the expected frequency is insufficient, Fisher's Exact test. For measurements repeated over time (e.g., postoperative pain scores, analgesic consumption, etc.), Repeated Measures ANOVA or, in the case of non-parametric measurements, the Friedman test will be used.

The study will include ASA 1-2 volunteer male and female patients over 18 years of age who will undergo elective septorhinoplasty surgery. Inclusion criteria:

* Septorhinoplasty surgery
* ASA 1-2 patients
* Men and women aged 18-65
* Informed consent and agreement to participate in the study Exclusion criteria: - ASA 3-4 and under 18 years of age
* Patients with serious renal, hepatological, cardiovascular, and pulmonary system diseases
* Patients allergic to paracetamol or ibuprofen
* Patients with bleeding diathesis, platelet dysfunction, gastrointestinal disease, peptic ulcer, pregnancy, planning pregnancy, and breastfeeding mothers
* Patients with ASA and those using anticoagulants Patients included in our study will be randomly assigned to three groups based on the preemptively administered medication using a computer-assisted randomization system by a blind investigator.

Patients participating in the study will be taken to the operating room 30 minutes prior to surgery with preemptive analgesic administration (SF, paracetamol, or ibuprofen). Routine monitoring procedures (pulse, ECG, SPO2, blood pressure, temperature, and ANI) will be performed. Routine anesthesia induction and maintenance will be carried out during the operation. Patients will be closely monitored throughout the case; operation time, complications, amount of opioid administered (µg/kg), and total opioid consumption will be recorded. In the postoperative period, patients will again have their pain monitored for 24 hours with patient-controlled intravenous (IV) PCA. Whether the patient needed opioid pain relief within 24 hours, and if so, when the first pain relief was needed, the number of times the patient-controlled IV PCA was administered, and the total amount of opioid used will be noted. Pain monitoring will be assessed using the NRS score in two separate ways: at 0, 1, 6, 12, and 24 hours postoperatively, at rest, and during activity (coughing and deep breathing). In addition, all patients will complete a postoperative QR-15 questionnaire to assess their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Septorhinoplasty surgery
* ASA1-2 patients
* Men and women aged 18-65
* Informed consent and acceptance to participate in the study

Exclusion Criteria:

* ASA 3-4 and under 18 years of age
* Patients with serious renal, hepatological, cardiovascular, or pulmonary system diseases
* Allergy to paracetamol or ibuprofen
* Patients with bleeding diathesis, platelet dysfunction, GI disease, peptic ulcers, pregnancy, planning pregnancy, and breastfeeding mothers
* Patients using ASA or anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS UNDERGOING SEPTORINOPLASTY SURGERY
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
ANALGESIA | 24 HOURS
  24-HOUR CUMULATIVE OPIOID CONSUMPTION
COMPILATION | POSTOPERATIVE 24TH HOUR
  POSTOPERATIVE QUALITY OF RECOVERY-15 SCALE
PAIN SCORE | 24 HOURS
  PAIN WILL BE ASSESSED POSTOPERATIVELY AT 0, 1, 6, 12, and 24 HOURS, BOTH AT REST AND DURING ACTIVITY (COUGHING AND DEEP BREATHING), USING THE NRS (Numeric Rating Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Cetinkaya, M.D., Principal Investigator — Samsun University Samsun Educational and Research Hospital
Locations (1):
- Samsun University Samsun Training and Research Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alshehri AA. Comparative Evaluation of Postoperative Pain Scores and Opioid Consumption in Septorhinoplasty After Administration of Single-Dose Preemptive Paracetamol and Ibuprofen: A Randomized Controlled Trial. Int Arch Otorhinolaryngol. 2023 Aug 4;27(3):e471-e477. doi: 10.1055/s-0042-1749386. eCollection 2023 Jul. PMID 37564463